CLINICAL TRIAL: NCT06691334
Title: Platelet Rich Plasma (PRP) and High Intensity Focused Ultrasound (HIFU) in Management of Stress Urinary Incontinence
Brief Title: Platelet Rich Plasma (PRP) and High Intensity Focused Ultrasound (HIFU) in Management of Stress Urinary Incontinence (SUI): Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Dina Mohamed Ahmed Srour, Doctor, Ain Shams Maternity Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Urinary incontinence
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: 10 cases will be group which is PRP injection 2 ml below urethra in one month interval. (Active Comparator): Procedure: PRP injection of 2ml platelet-rich plasma from centrifuged for 5 min patient's blood under urethra.
  Interventions: Device: PRP injection
- Group B: 10 cases will be group B which is PRP combined together with vaginal HIFU. (Active Comparator): Procedure: 3 cycles of vaginal HIFU together with 3 cycles of platelet-rich plasma injection treatment in 4 weeks intervals
  Interventions: Device: Hifu procedure and PRP injection

INTERVENTIONS:
Device: PRP injection — Active comparator: PRP 3 cycles of platelet-rich plasma injection treatment in 4 weeks intervals. Procedure: PRP injection of 2ml platelet-rich plasma from centrifuged for 5 min patient's blood under the urethra. Cycle patient will examined and asked to fill daily micturition plan International consolation on incontinence questionnaire-urinary incontinence short form (ICIQ UI SF), urogenital distress inventory (UDI-6), incontinence impact questionnaire (11Q-7) and over active bladder symptoms scores (OABSS).
  Arms: Group A: 10 cases will be group which is PRP injection 2 ml below urethra in one month interval.
Device: Hifu procedure and PRP injection — Procedure: PRP injection of 2ml platelet-rich plasma from centrifuged for 5 min patient's blood under urethra.And intravaginal Hifu in4 weeks intervals. Cycle patient will examined and asked to fill daily micturition plan International consolation on incontinence questionnaire-urinary incontinence short form (ICIQ UI SF), urogenital distress inventory (UDI-6), incontinence impact questionnaire (11Q-7) and over active bladder symptoms scores (OABSS).
  Arms: Group B: 10 cases will be group B which is PRP combined together with vaginal HIFU.

SUMMARY:
Previous studies Results show (PRP) is safe and effective in treating SUI, other studies show the result of energy base devices (Co2 laser, HIFU) are effective in treating of SUI .

This study add the effect both HIFU and PRP together in treating SUI.

DETAILED DESCRIPTION:
What is stress urinary incontinence (SUI)? Stress urinary incontinence (SUI) is when urine leaks out with sudden pressure on the bladder and urethra, causing the sphincter muscles to open briefly. With mild SUI, pressure may be from sudden forceful activities, like exercise, sneezing, laughing or coughing. If your SUI is more severe, you may also leak with less forceful activities like standing up, walking or bending over. Urinary "accidents" like this can range from a few drops of urine to enough to soak through the clothes SUI is a very common bladder problem for women. Key SUI statics About half of women age 65 and above find that they sometimes leak urine. How can SUI Affect life? Many people find that SUI gets in the way of daily and social activities. It can affect family and sexual relationships. Some people even begin to feel isolated and hopeless because of it The pelvic floor supports the bladder and urethra. If this area gets stretched, weakened or damaged, then SUI can happen. Pregnancy and childbirth can cause this.

PRP is extremely rich in growth factors and cytokines which regulate tissue reconstruction, PRP is an easily procedure and relatively inexpensive biological material, it is produce directly from patient blood and inject PRP under urethra to restore bulbourethral ligment .

HIFU is an energy-based medical technology with many clinical applications, a device is a non-invasive procedure that provides collagen remodeling and synthesis that may repair and restore pelvic floor and pubourethral ligment, it is non-invasive therapeutic technique, that uses non-ionized ultrasonic waves that provides collagen that tight the endopelvic fascia and adjacent tissues .

ELIGIBILITY:
Inclusion criteria:

* Women complain of SUI is the symptom of urinary leakage due to increased abdominal pressure, which can be caused by activities such as sneezing, coughing, exercise, lifting, and position change (American Urological Association 2017).
* Positive cough test when filled urinary bladder.
* Women chose non-invasive management rather than surgical management. • • Among the 20 patients enrolled, the average age was 30-60 years old.
* Urodynamic study proven the diagnosis.

Exclusion Criteria:

* Patient of previous operation or radiation
* Uncontrolled diabetes Neuromuscular disorder
* Uncontrolled psychiatric diseases
* Pregnancy
* Lactation
* Virgin
* Sepsis
* Active carcinoma
* Cystocele.
* Antiplatelet drug intake less than 7 days before and after procedure. - bleeding disorder.
* Patients cannot deal with Questionnaires.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
After one month of first session, the rate of Improvement of the stress urinary incontinence increased . | One month after first session
  Self-reported questionnaires were used to measure pre-Treatment symptom severity and post treatment symptom and severity.

SECONDARY OUTCOMES:
one month after complete three sessions ,the rate of Improvement of the urinary incontinence increased. | One month after complete three sessions
  Self-reported questionnaires were used to measure pre-Treatment symptom severity and post treatment symptom and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Srour, MS, Study Director — Ain Shams Maternity Hospital Egypt Ain Shams University Maternity Hospital
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt